CLINICAL TRIAL: NCT05308251
Title: Comparison of Hernia Sac Ligation Versus Invagination in Lichtenstein Tension Free Mesh Hernioplasty. Does Type of Hernia Have a Role on Outcomes?
Brief Title: Comparison of Hernia Sac Ligation Versus Invagination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Burak Ciftci, Principal Investigator, Samsun Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SamsunERH2020
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Hernia, Inguinal; Postoperative Pain; Recurrence
Keywords: indirect hernia sac; ligation; invagination
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Recurrence; Intussusception

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high ligation (Active Comparator): High ligation of the indirect hernia sac is traditional in inguinal hernia repairs. In this arm, patients with indirect inguinal hernia undergoing open mesh herniorrhaphy will have their hernia sac was opened and high ligated.
  Interventions: Procedure: Lichtenstein Mesh Hernioplasty
- non-ligation (Experimental): In this arm, the patients' hernia sac will be dissected high but not opened or ligated. The sac will be invaginated to the abdomen.
  Interventions: Procedure: Lichtenstein Mesh Hernioplasty

INTERVENTIONS:
Procedure: Lichtenstein Mesh Hernioplasty — The inguinal canal was opened and the hernia sac was dissected from the spermatic cord The deep inguinal ring was tightened with one or two polypropylene 2/0 sutures. The posterior wall of the inguinal canal was supported using the standard polypropylene mesh and fixed with 2/0 polyproline. The ilioinguinal nerve, iliohypogastric nerve, and genital branch of the genitofemoral nerve were preserved and care was taken to prevent entrapment.

SUMMARY:
Management of indirect hernial sac in inguinal hernia repairs has long been a subject of debate among general surgeons. Although hernial sac high ligation (HL) is a time-honored concept in groin hernia surgery, non-ligation/invagination is gaining more popularity. The aim of this study is to compare the effects of hernia sac ligation and invagination in patients with Lichtenstein mesh hernioplasty (LMH). Also, investigators aimed to investigate the possible association between the hernial defect size and postoperative early pain in both groups.

ELIGIBILITY:
Inclusion Criteria:

* unilateral uncomplicated indirect hernia
* elective operations
* spinal anesthesia

Exclusion Criteria:

* Bilateral hernias
* recurrent cases
* femoral-scrotal hernias
* those who refused to give consent
* those who were given general anesthesia besides spinal anesthesia
* those who were repaired with a method other than Lichtenstein mesh hernioplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain levels | postoperative period before discharge-1 year after discharge
  10-point Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
postoperative complications | postoperative period before discharge (mainly the first 24 hours)
  hematoma, seroma, wound infection, urinary retention
perioperative outcomes | postoperative period before discharge (mainly the first 24 hours)
  operative time (minutes), hospital stay (days)
recurrence | postoperative 1 year
  Number of patients with hernia recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Burak Ciftci, Principal Investigator — Samsun Education and Research Hospital
Locations (1):
- Samsun Eğitim ve Araştırma Hastanesi, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] HerniaSurge Group. International guidelines for groin hernia management. Hernia. 2018 Feb;22(1):1-165. doi: 10.1007/s10029-017-1668-x. Epub 2018 Jan 12. PMID 29330835
- [Result] Chen DC, Morrison J. State of the art: open mesh-based inguinal hernia repair. Hernia. 2019 Jun;23(3):485-492. doi: 10.1007/s10029-019-01983-z. Epub 2019 Jun 4. PMID 31165300
- [Result] Stylianidis G, Haapamaki MM, Sund M, Nilsson E, Nordin P. Management of the hernial sac in inguinal hernia repair. Br J Surg. 2010 Mar;97(3):415-9. doi: 10.1002/bjs.6890. PMID 20104504
- [Result] Delikoukos S, Lavant L, Hlias G, Palogos K, Gikas D. The role of hernia sac ligation in postoperative pain in patients with elective tension-free indirect inguinal hernia repair: a prospective randomized study. Hernia. 2007 Oct;11(5):425-8. doi: 10.1007/s10029-007-0249-9. Epub 2007 Jun 27. PMID 17594052
- [Result] Othman I, Hady HA. Hernia sac of indirect inguinal hernia: invagination, excision, or ligation? Hernia. 2014 Apr;18(2):199-204. doi: 10.1007/s10029-013-1081-z. Epub 2013 Apr 2. PMID 23546863
- [Derived] Ciftci AB, Ocak S. A comparison of hernia sac ligation versus invagination in Lichtenstein tension-free mesh hernioplasty: does the type of hernia play a role in outcomes? Hernia. 2022 Aug;26(4):1153-1159. doi: 10.1007/s10029-022-02637-3. Epub 2022 Jun 20. PMID 35725851